CLINICAL TRIAL: NCT05359081
Title: A 52-week, Open-label Study to Evaluate the Long-term Safety and Tolerability of SEP-363856 in Patients With Schizophrenia in Japan
Brief Title: A Clinical Trial to Evaluate the Long-term Safety and Tolerability of SEP-363856 in Patients With Schizophrenia in Japan
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Due to company business strategy
Sponsor: Sumitomo Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DA801202
Record Dates: First submitted 2022-04-27; First posted 2022-05-03 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2024-04

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — SEP-363856

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- SEP-363856 (Experimental): SEP-363856 (50 or 75 mg/day, flexible dose)
  Interventions: Drug: SEP-363856

INTERVENTIONS:
Drug: SEP-363856 — SEP-363856 50 mg or 75 mg, flexibly dosed once daily tablet for 52 weeks

SUMMARY:
A clinical study to investigate the long-term safety and torelability of SEP-363856 in clinically stable adult patients with schizophrenia in Japan.

DETAILED DESCRIPTION:
A phase 3, 52-week, open-label study to evaluate the long-term safety and tolerability of SEP-363856 in patients with schizophrenia in Japan. Participants will take flexible dose of SEP-363856 (50 mg/day and 75 mg/day) every night at bedtime for 52 weeks in an open-label manner.

ELIGIBILITY:
Inclusion Criteria:

1. Must be fully informed of and understand the objectives, procedures, and possible benefits and risks of the study, and give written informed consent prior to performing any study related activities.
2. Male or female between 18 to 65 years of age (inclusive) at the time of consent.
3. Must meet DSM 5 criteria for schizophrenia as established by clinical interview at Screening
4. Must have a PANSS total score >=60 at Screening and Baseline.
5. Must have a CGI-S score >=3 at Screening and Baseline
6. Judged to be clinically stable (i.e., no evidence of an acute exacerbation) by the Investigator for at least 8 weeks prior to Baseline and has had no change in antipsychotic medication(s) (minor dose adjustments for tolerability purposes are permitted) for at least 6 weeks prior to Screening
7. In the opinion of the Investigator, subjects must be generally healthy based on Screening medical history, physical examination, vital signs, ECG, and clinical laboratory values (hematology, chemistry, and urinalysis).

Exclusion Criteria:

1. Have a DSM-5 diagnosis or presence of symptoms consistent with a DSM-5 diagnosis other than schizophrenia. Exclusionary disorders include but are not limited to alcohol use disorder or substance (other than nicotine or caffeine) use disorder within past 12 months or for a total of >= 10 years during the subject's lifetime, major depressive disorder, bipolar I or II disorder, schizoaffective disorder, obsessive compulsive disorder, and posttraumatic stress disorder. Symptoms of mild to moderate mood dysphoria or anxiety are allowed so long as these symptoms have not been a focus of primary treatment
2. At significant risk of harming self, others, or objects based on Investigator's judgment.
3. Have any clinically significant unstable medical condition or any clinically significant chronic disease that in the opinion of the Investigator, would limit the subject's ability to complete and/or participate in the study.
4. Female subjects who are pregnant or lactating.
5. Have any clinically significant abnormal laboratory value(s) at Screening (hematology, chemistry, and urinalysis) as determined by the Investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2022-05-16 (Actual); Primary Completion 2024-03-21 (Actual); Study Completion 2024-03-28 (Actual)

PRIMARY OUTCOMES:
The incidence of overall adverse events (AEs), serious adverse events (SAEs), and AEs leading to discontinuation. | Week 52
  Evaluate the long-term safety and tolerability of flexible dosed SEP-363856 (50 and 75 mg/day) in subjects with schizophrenia by the incidence of overall adverse events (AEs), serious AEs (SAEs), and AEs leading to discontinuation.

CONTACTS AND LOCATIONS:
Locations (51):
- Japan (51):
  - Hotei Hospital, Konan-shi, Aichi-ken
  - Heart Care Clinic Omachi, Akita, Akita
  - Seinan Hospital, Hachinohe-shi, Aomori
  - Ishigooka Hospital, Chiba, Chiba
  - Kohnodai Hospital National Center for Global Health and Medicine, Ichikawa-shi, Chiba
  - Fukui Hospital, Fukui-shi, Fukui
  - Ai Sakura Clinic, Fukuoka, Fukuoka
  - Inokuchi Noma Hospital, Fukuoka, Fukuoka
  - Kuramitsu Hospital, Fukuoka, Fukuoka
  - Medical corporation Shinseikai Kaku Mental Clinic, Fukuoka, Fukuoka
  - Mental Clinic Sakurazaka, Fukuoka, Fukuoka
  - Shiranui Hospital, Omuta-shi, Fukuoka
  - Takeda General Hospital, Aizuwakamatsu-shi, Fukushima
  - Medical Corporation Kishikai Kishi Hospital, Kiryu-shi, Gunma
  - Hayakawa Clinic, Kure-shi, Hiroshima
  - NHO Kure Medical Center and Chugoku Cancer Center, Kure-shi, Hiroshima
  - Goryokai Hospital, Sapporo, Hokkaido
  - Tatsuta Clinic, Chuo-ku, Kobe-shi, Hyōgo
  - Kishiro Mental Clinic, Kawasaki-shi, Kanagawa
  - Musashikosugi J Kokorono Clinic, Kawasaki-shi, Kanagawa
  - Hino Hospital, Yokohama, Kanagawa
  - Miki Mental Clinic, Yokohama, Kanagawa
  - Yamatenomori Kokorono Clinic, Yokohama, Kanagawa
  - Tosa Hospital, Kochi, Kochi
  - Kouyoudai Hospital, Kumamoto, Kumamoto
  - Satokai Yuge Hospital, Kumamoto, Kumamoto
  - Miyazaki Prefectural Miyazaki Hospital, Miyazaki, Miyazaki
  - Ozawa Mental Clinic, Matsumoto-shi, Nagano
  - Okayama Psychiatric Medical Center, Okayama, Okayama-ken
  - NHO Ryukyu Hospital, Kunigami-gun, Okinawa
  - Akari Clinic, Naha, Okinawa
  - Miebashi Clinic, Naha, Okinawa
  - Barclay Imuro Mental Clinic, Urasoe-shi, Okinawa
  - Shiroma Clinic, Urasoe-shi, Okinawa
  - Kansai Medical University Medical Center, Moriguchi-shi, Osaka
  - Keihan Hospital, Moriguchi-shi, Osaka
  - NHO Hizen Psychiatric Center, Kanzaki-gun, Saga-ken
  - Rainbow & Sea Hospital, Karatsu-shi, Saga-ken
  - Inuo Mental Care Hospital, Tosu-shi, Saga-ken
  - Nishi Kumagaya Hospital, Kumagaya-shi, Saitama
  - Mental Clinic Minami, Saitama-shi, Saitama
  - Ryokuwakai Stresscare Hibiya Clinic, Chiyoda-ku, Tokyo
  - Murakami Hospital, Edogawa-ku, Tokyo
  - Narimasu Kosei Hospital, Itabashi-ku, Tokyo
  - Senzoku Psychosomatic Medicine Clinic, Meguro-ku, Tokyo
  - Sakura-shinmachi Mental Clinic, Setagaya-ku, Tokyo
  - Sangenjaya Neurology- Psychosomatic Clinic, Setagaya-ku, Tokyo
  - Sangubashi Kokorono Clinic, Shibuya-ku, Tokyo
  - Ohwa Mental Clinic, Toshima-ku, Tokyo
  - Sanyo Hospital, Sakata-shi, Yamagata
  - Yamagata Sakuracho Hospital, Yamagata, Yamagata

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Halff EF, Rutigliano G, Garcia-Hidalgo A, Howes OD. Trace amine-associated receptor 1 (TAAR1) agonism as a new treatment strategy for schizophrenia and related disorders. Trends Neurosci. 2023 Jan;46(1):60-74. doi: 10.1016/j.tins.2022.10.010. Epub 2022 Nov 8. PMID 36369028